CLINICAL TRIAL: NCT06179511
Title: A Modular Phase I/II, Open-label, Multicenter Study to Assess the Safety, Tolerability, Pharmacokinetics and Preliminary Antitumor Activity of AZD9829 as Monotherapy or in Combination in Patients With CD123-Positive Hematological Malignancies
Brief Title: Study of AZD9829 in CD123+ Hematological Malignancies
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: D9470C00001
Record Dates: First submitted 2023-10-27; First posted 2023-12-22 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Hematological Malignancies
Keywords: AZD9829; Anti-cancer agents; Dose escalation
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Module 1: Dose Escalation (Experimental): Ascending dose level cohorts of AZD9829 in AML and MDS participants.
  Interventions: Drug: AZD9829
- Module 1: Dose Optimization (Experimental): Characterizing the safety, tolerability, PK/PD, and preliminary antitumor activity of AZD9829 in CD123+ R/R AML participants, based on the data collected during dose escalation, dose optimization and backfill.
  Interventions: Drug: AZD9829

INTERVENTIONS:
Drug: AZD9829 — AZD9829 will be administered by IV infusion
  Arms: Module 1: Dose Escalation
Drug: AZD9829 — AZD9829 will be administered by IV infusion
  Arms: Module 1: Dose Optimization

SUMMARY:
This is a modular, multicentre, open-label, Phase I/II, dose-setting study. AZD9829 will be administered intravenously as monotherapy or in combination in participants with CD123 positive hematological malignancies.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age;
* CD123+ hematologic malignancy based on flow cytometry or immunohistochemistry by local laboratory;

  * R/R AML (except APL);
  * R/R HR-MDS with ≥5% bone marrow blast at time of inclusion;
* Had at least 1 prior line of therapy at currents histology, and have no available treatment options;
* ECOG performance status of ≤ 2.

The above is a summary, other inclusion criteria details may apply.

Exclusion Criteria:

* Active CNS leukemia;
* Previous treatment with any CD123 targeting therapy;
* Prior allogeneic HSCT, within 90 or cell therapy within 60 of start of therapy;
* Active GVHD that requires immunosuppressive treatment within 4 weeks prior to start of AZD9829;
* History of other malignancy(with certain exceptions);
* Active and uncontrolled infections;
* Unresolved AEs ≥2 Grade, from prior therapies.

The above is a summary, other exclusion criteria details may apply .

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2024-01-31 (Actual); Primary Completion 2025-10-31 (Actual); Study Completion 2026-03-23 (Estimated)

PRIMARY OUTCOMES:
Frequency of dose limiting toxicities (DLTs). | Module 1 - 28 days.
  DLTs are dose-limiting toxicities as defined in the study protocol.
Safety evaluation of AZD9829: Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | Module 1 - From informed consent until 60 days after last dose of AZD9829.
  Frequency, severity and relationship to study drug of AEs and SAEs
Identify RP2D in R/R AML patients. | Moldule 1 -From informed consent until 60 days after last dose of AZD9829.
  Incidence of AEs/SAEs and PK data

SECONDARY OUTCOMES:
Pharmacokinetics of AZD9829: Plasma Concentration of total antibody | Module 1 - From date of first dose of AZD9829 up until 30 days post last dose.
  Measurement of plasma concentration of conjugated and unconjugated antibody
Pharmacokinetics of AZD9829: Plasma Concentration of total unconjugated warhead | Module 1 - From date of first dose of AZD9829 up until 30 days post last dose.
  Measurement of plasma concentration of total unconjugated warhead
Pharmacokinetics of AZD9829: Area under the concentration time curve (AUC). | Module 1 - From date of first dose of AZD9829up until 30 days post last dose.
  Area under the plasma concentration-time curve.
Pharmacokinetics of AZD9829: Maximum plasma concentration of the study drug (Cmax). | Module 1 - From date of first dose of AZD9829 up until 30 days post last dose.
  Maximum observed plasma concentration of AZD9829.
Pharmacokinetics of AZD9829: Time to maximum concentration (tmax) | Module 1 - From date of first dose of AZD9829 up until 30 days post last dose.
  Time to maximum observed plasma concentration of the study drug.
Pharmacokinetics of AZD9829: Clearance | Module 1 - From date of first dose of AZD9829 up until 30 days post last dose.
  The volume of plasma from which the study drug is completely removed per unit time.
Pharmacokinetics of AZD9829: Half-life (t 1/2) | Module 1 - From date of first dose of AZD9829 up until 30 days post last dose.
  Terminal elimination half-life.
Pharmacokinetics of AZD9829: Anti-Drug Antibodies (ADA) | Module 1 - From date of first dose of AZD9829 up until 30 days post last dose.
  Evaluating the number of patients who develop anti-drug antibodies (ADA) during treatment.
Pharmacokinetics of AZD9829: Anti-Drug Antibodies (ADA) | Module 1 - From date of first dose of AZD9829 up until 30 days post last dose.
  Evaluating the percentage of patients who develop anti-drug antibodies (ADA) during treatment.
To determine the immunogenicity of AZD9829. | Module 1 - From first dose to the 30-Day SFU visit
  The number of participants who develop ADA (Anti Drug Antibodies).
To determine the immunogenicity of AZD9829. | Module 1 - From first dose to the 30-Day SFU visit
  The percentage of participants who develop ADA (Anti Drug Antibodies).
Overall Response Rate (ORR) | Module 1 - From first dose of AZD9829 until disease progression or end of the study (upto approximately 1 year)
  Overall response rate disease assessments in accordance with ELN2022 recommendations for AML and IWG 2006/2018 for MDS.
Composite Complete Response Rate (CCRR) | Module 1 - From first dose of AZD9829 up to approximately 1 year.
  Composite CR rate disease assessment in accordance with ELN2022 for AML and IWG 2006/2018 for MDS.
Complete remission with incomplete hematologic recovery (CRi) | Module 1 - From first dose of AZD9829 up to approximately 1 year.
  The endpoint of complete remission with CRi as defined by ELN2022 criteria.
Complete Response (CR) | Module 1 - From first dose of AZD9829 up to approximately 1 year.
  Complete response (CR) according to ELN2022 for AML and IWG 2006/2018 for MDS.
Duration of Response (DoR) | Module 1 -Time from first documented response until disease progression or death (approximately 1 year).
  Time from first documented response until the date of relapse or death.
Time to Response (TTR) | Module 1 - From first dose of AZD9829 until complete remission, disease progression or death (approximately 1 year).
  Time from first dose to the achievement of first overall response. Disease assessments will follow ELN2022 for AML and IWG 2006/2018 for MDS.
Time to Next Treatment (TTNT) | Module 1 - From first dose of AZD9829 until the date of subsequent anti-leukemia-therapy or death (approximately 1 year).
  The time from the start of treatment date until the date of subsequent antileukemia therapy.
Progression-free Survival (PFS) | Module 1 - From first dose of AZD9829 until disease progression or death (approximately 1 year).
  The time from the start of treatment date until the date of disease progression or death.
Overall Survival (OS) | Module 1 - From first dose of AZD9829 until death (approximately 1 year).
  The time from the start of treatment date until death.
Event-free Survival (EFS) | Module 1 - From first dose of AZD9829 until disease progression, death, or initiation of a new anti-leukemic therapy (approximately 1 year).
  The time from the start of treatment date to disease progression, death, or initiation of a new anti-leukemic therapy.

CONTACTS AND LOCATIONS:
Locations (21):
- United States (7):
  - Research Site, Duarte, California
  - Research Site, St Louis, Missouri
  - Research Site, New York, New York
  - Research Site, Chapel Hill, North Carolina
  - Research Site, Columbus, Ohio
  - Research Site, Houston, Texas
  - Research Site, Milwaukee, Wisconsin
- Australia (2):
  - Research Site, Heidelberg
  - Research Site, Melbourne
- Research Site, Tianjin, China
- Research Site, Frankfurt, Germany
- Research Site, Bologna, Italy
- Japan (3):
  - Research Site, Kashiwa
  - Research Site, Osaka
  - Research Site, Yoshida-gun
- Research Site, Seoul, South Korea
- Spain (2):
  - Research Site, Barcelona
  - Research Site, Salamanca
- Taiwan (2):
  - Research Site, Tainan
  - Research Site, Taipei
- Research Site, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home